CLINICAL TRIAL: NCT07301814
Title: Clinical Application of PET Imaging Targeting CLDN18.2 in Malignant Tumors
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: XLan-0785
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer; Pancreatic Cancer; Cholangiocarcinoma Cancer; Esophageal Cancer
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Specific PET imaging agents targeting CLDN18.2 — The project aims to perform integrated PET/MR or PET/CT imaging in patients with histologically confirmed or clinically suspected gastric cancer, pancreatic cancer, cholangiocarcinoma, or other malignant tumors with high Claudin18.2 (CLDN18.2) expression, as well as healthy volunteers. This study utilizes a CLDN18.2-specific PET imaging probe (e.g., [^68Ga]Ga-labeled humanized antibody fragment) to evaluate the feasibility, accuracy, and clinical value of non-invasive, in vivo CLDN18.2 visualization.

SUMMARY:
The project aims to perform integrated PET/MR or PET/CT imaging in patients with histologically confirmed or clinically suspected gastric cancer, pancreatic cancer, cholangiocarcinoma, or other malignant tumors with high Claudin18.2 (CLDN18.2) expression, as well as healthy volunteers. This study utilizes a CLDN18.2-specific PET imaging probe (e.g., [^68Ga]Ga-labeled humanized antibody fragment) to evaluate the feasibility, accuracy, and clinical value of non-invasive, in vivo CLDN18.2 visualization.

For patients with malignant tumors, the study will assess the diagnostic performance of CLDN18.2-targeted PET in identifying tumor lesions, compare the imaging results with gold-standard histopathology, determine the location, extent, and metabolic features of CLDN18.2-positive lesions, and evaluate tumor burden and treatment stratification value compared with [^18F]FDG PET imaging. These results may assist in patient selection for CLDN18.2-targeted therapies (e.g., Zolbetuximab), guide clinical decision-making, and provide early prediction of therapeutic response.

For healthy volunteers, pharmacokinetic profiling will be conducted to investigate the biodistribution, clearance, and safety of the radiotracer in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Each participant must meet all inclusion criteria to be eligible to participate in the study:

  1. The participant or their legal representative is able to sign the informed consent form with signature and date;
  2. Commit to adhering to the research procedures and cooperating in the implementation of the entire research process;
  3. Adult patients or healthy volunteers (aged 18-70 years), male or female;
  4. Patients with malignant tumors such as gastric cancer, pancreatic cancer, bile duct cancer, esophageal cancer, etc., suspected or diagnosed clinically (supporting evidence includes serum tumor markers, ultrasound, CT, MRI, and other imaging data, as well as histopathological examination), and in good general condition;
  5. Meet specific laboratory test results;
  6. Women of childbearing age must use contraception for at least one month before screening and commit to using contraception throughout the study period and continuing it until the specified time after the study ends;
  7. Other set inclusion criteria.

Exclusion Criteria:

* All subjects who meet any exclusion criteria baseline will be excluded from the study:

  1. Those unable to complete PET/MR or PET/CT scans (including those unable to lie flat, claustrophobia, radiation phobia, etc.);
  2. Those with other comorbidities;
  3. Patients known to be allergic to the targeted CLDN18.2 PET imaging agent or synthetic excipients; fasting blood glucose level exceeding 11.0 mmol/L before injection of 18F-FDG;
  4. Those with a history of concomitant medication use;
  5. Patients considered to have poor compliance by the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or confirmed malignant tumors such as gastric adenocarcinoma, pancreatic cancer, bile duct cancer, esophageal adenocarcinoma, etc. (supporting evidence includes serum tumor markers, ultrasound, CT, MRI, and histopathological examination of tissue, etc.), and in good general condition.
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual and standardized uptake values assessment of lesions and biodistribution | 1 year
  At least two experienced nuclear medicine physicians will conduct a visual analysis using consensus reading. The standardized uptake value (SUV) of the tumor and organs will be measured after a semiquantitative analysis is performed for each case. The SUV ranges from 0 to infinity, and a higher score means a higher uptake of targeting CLDN18.2 nuclear probe by the tumor, which implies a greater threat of the tumor being malignant or a higher stage.

SECONDARY OUTCOMES:
Radioactivity in the blood and urine samples | 1 year
  Blood samples were collected at 25 minutes, 55 minutes and 115 minutes after injection.
Pathological sections of tumour tissue | 1 year
  The excised tumour tissue was taken for immunohistochemistry to verify its CLDN18.2 expression

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, PhD, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, China, Wuhan, Hubei, China